CLINICAL TRIAL: NCT00977145
Title: Evaluation of the Safety and Immunogenicity of Intratumoral Injection of Interferon Gamma During Vaccination in Patients With Subcutaneous or Cutaneous Metastases of Melanoma
Brief Title: Evaluating the Safety and the Biological Effects of Intratumoral Interferon Gamma and a Peptide-Based Vaccine in Patients With Melanoma
Acronym: Mel 51
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed short of the enrollment goal, due to slow enrollment and adequate data to address endpoints
Sponsor: Craig L Slingluff, Jr (Other)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14215
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Melanoma
Keywords: melanoma; peptide vaccine; interferon gamma; immunotherapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intratumoral IFN-gamma plus MELITAC 12.1, (Experimental): intratumoral IFN-gamma plus systemic vaccination with MELITAC 12.1, an emulsion of a mixture of 12 class I MHC-restricted melanoma-derived peptides (12-MP) and a class II MHC-restricted tetanus toxoid-derived helper peptide (Peptide-tet).
  Interventions: Biological: A combination of intratumoral IFN-gamma plus systemic vaccination with MELITAC 12.1

INTERVENTIONS:
Biological: A combination of intratumoral IFN-gamma plus systemic vaccination with MELITAC 12.1 — Vaccine regimen: The vaccines will be administered in two treatment cycles. During cycle one, three vaccines will be administered over a 3-week period on days 1, 8, 15. During cycle two, three vaccines will be administered over a 9-week period on days 24, 43, 64. All participants will receive 12-MP (100 mcg each peptide) plus Peptide-tet (Peptide-tet; 200 mcg) administered in Montanide ISA-51 VG adjuvant. The vaccine will be administered subcutaneously (1 ml) and intradermally (1ml) at a single vaccination site.
  Intratumoral Interferon regimen: On day 22, patients will have one or more tumor sites injected with 0.5-2 million IU of IFN-gamma each, with a maximum dose of 2 million IU of IFN-gamma administered per patient. The number of lesions that are injected will be dependent on the availability and size of the lesions.

SUMMARY:
The goals of this study are to evaluate 1) the safety of administration of intratumoral interferon gamma with a peptide-based vaccine, in patients with melanoma and 2) the biological effects of the vaccine. These include an examination of changes within the tumor following vaccination and the evaluation of T cell responses to the vaccine both in the blood and at the sight of tumor.

DETAILED DESCRIPTION:
Melanoma vaccines have been associated with major regressions in a small percentage of patients with advanced measurable disease. This provides proof-of-principle of the potential for clinical benefit with melanoma vaccines however, the current response rate is low. Thus, there is a critical need for additional new therapies for melanoma, both for adjuvant therapy of high-risk resected melanoma and for therapy of patients who are not candidates for, or fail, other therapies in the setting of advanced disease.

It is generally agreed that one mechanism to improve the immunologic outcomes of vaccine therapy is to optimize T cell trafficking to the tumor site. CXCR3 is the chemokine receptor on T cells which directs them to sites of inflammation by following the chemokine gradient. The ligands for CXCR3 (CXCL9 (MIG), CXCL10 (IP-10) and CXCL11 (I-TAC)) are known to be induced by interferon gamma. This protocol proposes administering a peptide vaccine to activate tumor antigen-specific CD8+ T cells expressing CXCR3, followed by intratumoral interferon gamma to increase CXCR3 ligands (CXCL9-11) at the tumor site and recruit the CXCR3+ T cells.

The primary goals of the proposed work are to assess the safety of the combination of peptide vaccine and intratumoral interferon gamma and to assess the immunologic outcomes at the tumor site.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with stage IIIB, IIIC or IV melanoma. Staging must be confirmed by cytological or histological examination. Staging of cutaneous melanoma will be based on the revised AJCC staging system.
2. Patients must have adequate cutaneous or subcutaneous metastases of melanoma readily accessible for biopsy to provide a minimum of 0.3 cm3 of tissue per biopsy (approximately 0.85 cm by 0.85 cm x 0.85 cm or five 2mm core biopsies) at each time point. Additionally, at least one of the subcutaneous or cutaneous metastases must be accessible to intratumoral IFN-gamma administration. Several scenarios may fulfill the tumor burden requirement. For example, a patient may have one large lesion from which core biopsies can be taken for the first and second biopsy time points and then the entire lesion excised for the final tissue sample. Alternatively, a patient may have three lesions, each ≥0.3 cm3, and these lesions would be excised sequentially as biopsies 1, 2 and 3. Other combinations are acceptable.

   The intent is to limit this study to patients with cutaneous or subcutaneous melanoma metastasis rather than lymph node metastasis. There may be cases where a subcutaneous nodule cannot be definitively characterized as a non-nodal metastasis at the start of the trial - these patients may be included.
3. Participants with ocular, mucosal or unknown primaries and participants with multiple primaries will be eligible.
4. Participants who have had brain metastases may be eligible in selected circumstances:

   Patients with less than or equal to 3 metastases may eligible as long as the following 3 criteria are true:
   * The brain metastases have been completely removed by surgery or have been treated completely by stereotactic radiotherapy. Stereotactic radiotherapy, such as gamma knife, can be used up to 1 week prior to study entry.
   * There has been no evident growth of any brain metastasis since treatment.
   * No metastasis greater than 2 cm at the time of protocol entry

   Patients with greater than 3 metastases may be eligible if the above 3 criteria are met and if at least one year has elapsed since the last treatment.
5. All participants must have:

   * ECOG performance status of 0 or 1
   * Ability and willingness to give informed consent
6. Laboratory parameters - The following laboratory parameters will be required for all participants. If a lab value appears to be an error or a result of a transient or treatable condition, the investigator will use his/her clinical judgment to decide if the test may be repeated. The requirements for inclusion are as follows:

   * HLA-A1, -A2, -A3, or -A11+
   * ANC > 1000/mm3
   * Platelets > 100,000/mm3
   * Hgb > 9 g/dL
   * HGBA1C < 7%
   * Hepatic:

     * AST and ALT ≤ 2.5 x upper limits of normal (ULN)
     * Bilirubin ≤ 2.5 x ULN
     * Alkaline phosphatase ≤ 2.5 x ULN
   * Renal

     o Creatinine ≤ 1.5 x ULN
   * Serology (within 6 months of study entry)

     * HIV negative
     * Hepatitis C negative
   * LDH up to 2 x ULN
7. Age 18 years or older at the time of trial entry
8. Participants must have at least one intact (undissected) axillary and/or inguinal lymph node basin

Exclusion Criteria:

1. Patients who have had brain metastases unless they meet the criteria outlined above in the inclusion criteria.
2. Patients who are currently receiving systemic cytotoxic chemotherapy, radiation, or other experimental therapy, or who have received this therapy within the preceding 4 weeks. Gamma knife or stereotactic radiosurgery may be administered within the prior 4 weeks, but must not be administered less than one week prior to study enrollment. Patients who are currently receiving nitrosoureas or who have received this therapy within the preceding 6 weeks.
3. Patients will not be eligible if there is clinically detectable melanoma deemed likely by the investigator to require intervention during the first 3 months of the study that would require premature discontinuation. Examples for such circumstances may include untreated bone metastases at risk for fracture, and rapidly progressive low volume disease.
4. Patients with known or suspected allergies to any component of the vaccine.
5. Patients receiving the following medications at study entry or within the preceding 4 weeks are excluded:

   * Agents with putative immunomodulating activity (with the exception of non-steroidal anti-inflammatory agents and topical steroids)
   * Allergy desensitization injections.
   * Systemic corticosteroids, administered parenterally or orally. Inhaled steroids (e.g. Advair®, Flovent®, Azmacort®) are not permitted. Topical corticosteroids are acceptable, including steroids with very low solubility administered nasally for local effects only (e.g. Nasonex®).
   * Any growth factors (e.g. GM-CSF, G-CSF, erythropoietin).
   * Interferon therapy
   * Interleukin-2 or other interleukins.
6. Prior melanoma vaccinations may be an exclusion criterion in some circumstances:

   * Patients who have recurred or progressed either after or during administration of a melanoma vaccine may be eligible to enroll 12 weeks following their last vaccination.
   * Patients may have been vaccinated previously with peptide vaccines (including MELITAC 12.1 and similar vaccines) or with non-peptide vaccines.
7. Other investigational drugs or investigational therapy if the patient is currently taking those drugs/therapy, or if they have received the drugs/therapy within 1 month.
8. Pregnancy or the possibility of becoming pregnant during vaccine administration. Female patients of child-bearing potential must have a negative pregnancy test (urinary or serum beta-HCG) prior to administration of the first vaccine dose. Males and females must agree, in the consent form, to use effective birth control methods during the course of vaccination. Women must also not be breast feeding. This is consistent with existing standards of practice for vaccine and chemotherapy protocols.
9. Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.
10. Patients classified according to the New York Heart Association classification as having Class III or IV heart disease.
11. Patients with a body weight < 110 lbs because of the amount and frequency with which blood will be drawn
12. Participants must not have had prior autoimmune disorders requiring cytotoxic or immunosuppressive therapy, or autoimmune disorders with visceral involvement. Participants with an active autoimmune disorder requiring these therapies are also excluded. The following will not be exclusionary:

    * The presence of laboratory evidence of autoimmune disease (e.g. positive ANA titer) without symptoms
    * Clinical evidence of vitiligo
    * Other forms of depigmenting illness
    * Mild arthritis requiring NSAID medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Safety: To determine the safety of administration of intratumoral interferon gamma with a peptide-based vaccine in patients with cutaneous or subcutaneous metastases of melanoma. | 6 months
Biologic effect: To evaluate the biological effects of vaccine plus IFN-gamma at the tumor site, to include expression of CXCR3 ligands (CXCL9, CXCL10 & CXCL11) and the magnitude of infiltration of CD8+ CXCR3+ T cells and vaccine-specific T cells. | 6 months

SECONDARY OUTCOMES:
To estimate the effects of vaccine on CXCR3 expression by circulating antigen-experienced CD4 and CD8 T cells. | 6 months
To estimate the effects of vaccine plus IFN-gamma on changes in the percentage of FoxP3+ CD25hi CD4+ (putative regulatory T cells, T regulatory cells) among tumor infiltrating T cells. | 6 months
To obtain preliminary data on the variability of immunologic parameters among multiple biopsies of subcutaneous or cutaneous metastases of melanoma. | 6 months
To obtain preliminary data on the clinical response of cutaneous or subcutaneous metastases of melanoma to the proposed combination regimen. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Tran CA, Lynch KT, Meneveau MO, Katyal P, Olson WC, Slingluff CL Jr. Intratumoral IFN-gamma or topical TLR7 agonist promotes infiltration of melanoma metastases by T lymphocytes expanded in the blood after cancer vaccine. J Immunother Cancer. 2023 Feb;11(2):e005952. doi: 10.1136/jitc-2022-005952. PMID 36746511